CLINICAL TRIAL: NCT03718169
Title: Using a Smartphone Application to Deliver a Gender-specific Smoking Cessation Programme Among Female Smokers in Hong Kong
Brief Title: Smartphone Application-based Smoking Cessation Programme Among Female Smokers
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. LI William Ho Cheung, Associate Professor, The University of Hong Kong
Other Study IDs: KE funding
Record Dates: First submitted 2018-08-26; First posted 2018-10-24 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-06

CONDITIONS: Smoking Cessation
Keywords: women
MeSH Terms: conditions — Smoking Cessation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hong Kong female smokers: Hong Kong female smokers will be invited to fill in questionnaires about their current smoking situation and quit intention.
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires — Female smokers will be asked to complete a structured questionnaire at smoking hotspots. In addition, the smokers will respond to the same questionnaire at 6 months via telephone. The structured questionnaire will collect information related to their demographic characteristics and quitting behaviors, i.e. self-reported abstinence, smoking reduction and quit attempts.

SUMMARY:
This project aims to develop a smartphone application to deliver a gender-specific programme for female smokers in Hong Kong. Through the smartphone application, we expect that our gender-specific smoking cessation programme can reach more female smokers in Hong Kong. The objectives is to promote smoking cessation among female smokers in Hong Kong.

DETAILED DESCRIPTION:
This is a one-year project, and it will be divided into 2 Phases. Phase I will focus on translating our gender-specific smoking cessation programme into a smartphone application. In Phase II, the investigators will promote the smartphone application to female smokers in the community.

Phase I: Translating our gender-specific smoking cessation programme into a smartphone application To translate our gender-specific smoking cessation programme into a smartphone application, an expert panel will be formed. The panel members include a chair professor, an associate professor, an assistant professor, a research assistant professor and a postdoctoral fellow, with all of whom have considerable experience in conducting studies on smoking cessation and tobacco control. The content of the smartphone application will be designed according to the gender-specific smoking cessation programme delivered by our women Quitline. In particular, the smartphone application aims to help female smokers abstain from cigarettes by their readiness to quit. For female smokers who are in the pre-contemplation or contemplation stage, the smartphone application will motivate them to quit by instructing them to list out the reasons for quitting, and providing them information about the damaging effects of smoking on health, especially those are specific to women. Regarding female smokers in the preparation stage, the smartphone application will assist them to individualize their own quit plan by computerized instructions, and provide generic tips how they can achieve abstinence step-by-step. Concerning female smokers in the action stage, skills for overcoming cigarette craving and withdrawal symptoms will be presented. In addition, hazardous effects of smoking will pop-up in their smartphones to remind them of smoking cessation throughout their quitting process. To address the needs and concerns of female smokers, gender-specific elements have been integrated into the smartphone application. In particular, the smartphone application will correct their misconceptions that smoking can be a method to control body weight and manage stress. At the same time, the smartphone application will display information about proper weight-loss strategies and relaxation techniques. Female smokers who need more intensive counseling can also contact our Quitline via the smartphone application.

Phase II: Promoting the smartphone application for female smokers in the community In order to promote the smartphone application for female smokers, the investigators plan to recruit 30 students from the University of Hong Kong to join this project. All recruited students will be invited to participate in a 1-day training workshop organized by our team. During the training workshop, the students will be educated on smoking hazards, the basic principles of smoking cessation and tobacco control policies.

Female smokers will be recruited in smoking hotspots where rubbish bins with a collector of cigarette butts are nearby. The trained university students will approach female smokers at the smoking hotspots, and deliver a small souvenir to them. The souvenir is a pack of tissue paper, with its packaging containing smoking cessation messages and the QR code of the smartphone application. If the smokers accept the souvenir, the students will then introduce this project. For female smokers who are interested to join, the students will assist them to download the smartphone application, briefly go through its content, and encourage them to use it. To remind the female smokers to continuously use the smartphone application for smoking cessation, warning messages about the hazardous effects of smoking will pop up weekly in their smartphones.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong female resident aged 18 or above
* Able to communicate in Chinese (Cantonese)
* Current Smokers

Exclusion Criteria:

* Have difficulty to communicate via telephone
* Having queries irrelevant to tobacco control

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only female smokers will be selected.
Study Population: Hong Kong female smokers.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
7-days point prevalence smoking abstinence at 6-month | 6-month follow-up
  7-days point prevalence smoking abstinence is measured at 6-month. A questionnaire asking smoking status, quitting experience and difficulty in quitting was designed to assess the self-reported smoking abstinence at 6-month.

SECONDARY OUTCOMES:
Bio-chemical validated smoking abstinence at 6-month | 6-month follow-up
  Bio-chemical validated smoking abstinence is measured at 6-month. The participants who claim to have quitted smoking for at least 7 days are invited for biochemical validation (measurement of saliva cotinine level and exhaled carbon monoxide level) at 6-month. The participants are need to get the results of CO≤ 4ppm, and continine level ≤30 ng/ml as passing results.

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Cheung Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No